CLINICAL TRIAL: NCT02105610
Title: Volatile Anesthetics to Reduce Mortality in Cardiac Surgery: A Multicentre Randomized Controlled Study
Brief Title: Volatile Anesthetics to Reduce Mortality in Cardiac Surgery
Acronym: MYRIAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Associate Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VOLATILE/38/OSR
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Aortocoronary Bypass; Cardiac Surgery; Coronary Artery Bypass Grafting
Keywords: volatile anesthetics; desflurane; isoflurane; sevoflurane; TIVA; cardiac surgery; mortality; anesthesia; intensive care
MeSH Terms: interventions — Desflurane; Isoflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- volatile anesthetics (desflurane, isoflurane, sevoflurane) (Experimental)
  Interventions: Drug: desflurane, isoflurane, sevoflurane
- total intravenous anesthesia (Active Comparator)
  Interventions: Drug: total intravenous anesthetics

INTERVENTIONS:
Drug: desflurane, isoflurane, sevoflurane
  Arms: volatile anesthetics (desflurane, isoflurane, sevoflurane)
Drug: total intravenous anesthetics
  Arms: total intravenous anesthesia

SUMMARY:
There is initial evidence that the choice of anesthesia can influence survival in the specific setting of coronary artery bypass grafting surgery (CABG).

A recent international consensus conference included volatile agents among the few drugs/techniques/strategies that might reduce perioperative mortality in cardiac surgery and that should be further studied. Volatile anesthetics (desflurane, isoflurane and sevoflurane) have non-anesthetic pharmacological characteristics that confer cardiac protection when compared to Total IntraVenous Anesthesia (TIVA). Several randomized controlled studies were summarized in a meta-analysis that documented a reduction in perioperative cardiac troponin release and mortality in patients receiving volatile anesthetics when compared to patients receiving a TIVA. There are four published studies (Bignami et al. 2009) (De Hert et al. 2009) (Jackobsen et al. 2007) (Landoni et al. 2007) suggesting that these benefits can translate into a reduced mortality rate in patients receiving volatile agents. The level of evidence for these four studies is not high (one meta-regression, one underpowered randomized controlled study, one retrospective study and one meta-analysis of small randomized studies) and there is need for a large multicentre randomized controlled study to confirm these findings, as suggested by the international consensus conference on this topic published in 2011 (Landoni et al 2011).

The purpose is to provide a large multicentre controlled randomized trial to demonstrate that volatile anesthetics can reduce 1 year mortality from 3% to 2% in patients undergoing CABG (either with or without cardiopulmonary bypass).

The results of this study can support the use of volatile agents in all CABG procedures worldwide (more than 500.000 per year) with 2.500 lives saved per year (in the hypothesis that nowadays half the procedures are performed with a TIVA and that 1 year mortality can be reduced from 3% to 2% using volatile agents).

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* written informed consent
* scheduled procedures
* planned isolated CABG (multiple bypass are allowed; planned combined intervention such as CABG plus valve surgery are not allowed

Exclusion Criteria:

* pregnancy
* planned valve surgery or surgery on the aorta
* planned locoregional anesthesia without general anesthesia
* unstable or ongoing angina
* recent (< 1 month) or ongoing acute myocardial infarction
* use of sulfonylurea, theophylline or allopurinol
* previous unusual response to an anesthetic agent
* inclusion in other randomised controlled studies in the previous 30 days
* any general anesthesia performed in the previous 30 days
* emergency operation (not scheduled)
* Kidney or liver transplant in medical history
* Liver cirrhosis (Child B or C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5400 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: alberto zangrillo, Prof, Study Chair — Vita-Salute University of Milano
Locations (36):
- Mohammed Bin Khalifa Bin Sulman Al-Khalifa Cardiac Center - Bahrain, Bahrein, Bahrain
- Brazil (2):
  - Hospital das Clínicas da Faculdade de Medicina da USP - Istituto do Coracao, São Paulo, Barazil
  - Dante Pazzanese Institute of Cardiology, São Paulo
- Heart Center Pontica, Burgas, Bulgaria
- China (4):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Wuhan Asia Heart Hospital, Hubei
  - 1st Affiliated Hospital of Fourth Military University, Xi'an
- University Hospital Dubrava, Dubrava, Croatia
- Czechia (2):
  - General University Hospital, Charles University, Prague, Czech Republic
  - Institute for Clinical and Experimental Medicine, Prague, Czech Republic
- Egypt (2):
  - Mansoura University hospitals, Egypt, Egypt
  - Faculty of Medicine - Zagazig University, Zagazig
- Italy (9):
  - Policlinico San Orsola-Malpighi, Bologna
  - Spedali Civili, Brescia
  - Policlinico Universitario Magna Graecia, Catanzaro
  - Ospedale San Raffaele di Milano, Italy, Milan
  - Humanitas, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Policlinico Universitario Campus Biomedico, Roma
  - AOU Città della Salute e della Scienza, Torino
- Malaysia (4):
  - Hospital Pulau Pinang, George Town, Malaysia
  - Hospital Serdang, Lumpur, Malaysia
  - University Malaya Medical Centre, Lumpur, Malaysia
  - Sarawak General Hospital, Sarawak, Malaysia
- Hospital Santa Maria, Lisbon, Portugal
- Russia (7):
  - Federal Centre for Cardiac Surgery, Astrakhan
  - Scientific Research Institute for Complex Issues of Cardiovascular Disease, Kemerovo
  - Moscow Clinical Regional Research Institute, Moscow
  - Negovskiy Reanimatology Research Institute, Moscow
  - State Research Institute of Circulation Pathology, Novosibirsk
  - Federal Almazov Medical Research Centre, Saint Petersburg
  - Ural Institute of Cardiology, Yekaterinburg
- King Abdullah Medical City - KAMC, Mecca, Saudi Arabia
- Institute of Cardiovascular Diseases "Dedinje", Belgrade, Serbia

REFERENCES:
- [Background] Landoni G, Greco T, Biondi-Zoccai G, Nigro Neto C, Febres D, Pintaudi M, Pasin L, Cabrini L, Finco G, Zangrillo A. Anaesthetic drugs and survival: a Bayesian network meta-analysis of randomized trials in cardiac surgery. Br J Anaesth. 2013 Dec;111(6):886-96. doi: 10.1093/bja/aet231. Epub 2013 Jul 12. PMID 23852263
- [Background] Landoni G, Rodseth RN, Santini F, Ponschab M, Ruggeri L, Szekely A, Pasero D, Augoustides JG, Del Sarto PA, Krzych LJ, Corcione A, Slullitel A, Cabrini L, Le Manach Y, Almeida RM, Bignami E, Biondi-Zoccai G, Bove T, Caramelli F, Cariello C, Carpanese A, Clarizia L, Comis M, Conte M, Covello RD, De Santis V, Feltracco P, Giordano G, Pittarello D, Gottin L, Guarracino F, Morelli A, Musu M, Pala G, Pasin L, Pezzoli I, Paternoster G, Remedi R, Roasio A, Zucchetti M, Petrini F, Finco G, Ranieri M, Zangrillo A. Randomized evidence for reduction of perioperative mortality. J Cardiothorac Vasc Anesth. 2012 Oct;26(5):764-72. doi: 10.1053/j.jvca.2012.04.018. Epub 2012 Jun 20. PMID 22726656
- [Background] Landoni G, Lomivorotov V, Pisano A, Nigro Neto C, Benedetto U, Biondi Zoccai G, Gemma M, Frassoni S, Agro FE, Baiocchi M, Barbosa Gomes Galas FR, Bautin A, Bradic N, Carollo C, Crescenzi G, Elnakera AM, El-Tahan MR, Fominskiy E, Farag AG, Gazivoda G, Gianni S, Grigoryev E, Guarracino F, Hanafi S, Huang W, Kunst G, Kunstyr J, Lei C, Lembo R, Li ZJ, Likhvantsev V, Lozovskiy A, Ma J, Monaco F, Navalesi P, Nazar B, Pasyuga V, Porteri E, Royse C, Ruggeri L, Riha H, Santos Silva F, Severi L, Shmyrev V, Uvaliev N, Wang CB, Wang CY, Winterton D, Yong CY, Yu J, Bellomo R, Zangrillo A. MortalitY in caRdIAc surgery (MYRIAD): A randomizeD controlled trial of volatile anesthetics. Rationale and design. Contemp Clin Trials. 2017 Aug;59:38-43. doi: 10.1016/j.cct.2017.05.011. Epub 2017 May 19. PMID 28533194
- [Derived] Lomivorotov V, Ruzankin PS, Lembo R, Tarasenko AS, Chernyavskiy A, Crivellari M, Monaco F, Ruggeri L, Pieri M, Lomivorotova L, Belletti A. Volatile versus Total Intravenous Anesthesia for Coronary Artery Bypass Graft Surgery: Analysis of 1586 MYRIAD Trial Patients Managed with the Same Perioperative Protocol. Rev Cardiovasc Med. 2022 Jul 21;23(8):265. doi: 10.31083/j.rcm2308265. eCollection 2022 Aug. PMID 39076624
- [Derived] Landoni G, Lomivorotov VV, Nigro Neto C, Monaco F, Pasyuga VV, Bradic N, Lembo R, Gazivoda G, Likhvantsev VV, Lei C, Lozovskiy A, Di Tomasso N, Bukamal NAR, Silva FS, Bautin AE, Ma J, Crivellari M, Farag AMGA, Uvaliev NS, Carollo C, Pieri M, Kunstyr J, Wang CY, Belletti A, Hajjar LA, Grigoryev EV, Agro FE, Riha H, El-Tahan MR, Scandroglio AM, Elnakera AM, Baiocchi M, Navalesi P, Shmyrev VA, Severi L, Hegazy MA, Crescenzi G, Ponomarev DN, Brazzi L, Arnoni R, Tarasov DG, Jovic M, Calabro MG, Bove T, Bellomo R, Zangrillo A; MYRIAD Study Group. Volatile Anesthetics versus Total Intravenous Anesthesia for Cardiac Surgery. N Engl J Med. 2019 Mar 28;380(13):1214-1225. doi: 10.1056/NEJMoa1816476. Epub 2019 Mar 19. PMID 30888743